CLINICAL TRIAL: NCT04305405
Title: An Open-label Study to Evaluate the Pharmacokinetics and Pharmacodynamics and Long-term Safety of Benralizumab Administered Subcutaneously in Children With Severe Eosinophilic Asthma
Brief Title: PK/PD and Long Term Safety Study of Benralizumab in Children With Severe Eosinophilic Asthma
Acronym: TATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Parexel (Industry); Covance (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D3250C00025
Record Dates: First submitted 2019-11-15; First posted 2020-03-12 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Severe Uncontrolled Asthma
Keywords: Pediatric; PK; severe asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): Below 35 kilos
  Interventions: Drug: Benralizumab
- Dose 2 (Experimental): Greater than/equal to 35 kilos
  Interventions: Drug: Benralizumab

INTERVENTIONS:
Drug: Benralizumab — Dose will be stratified by body weight at screening: Patients will receive Dose 1 or Dose 2 of Benralizumab administered by SC injection at Day 0 and Weeks 4, 8, and 16, 24, 32, and 40.

SUMMARY:
This study will evaluate the PK, PD and long-term safety of Benralizumab administered subcutaneously in 30 children aged 6 to 11 years with severe eosinophilic asthma. Up to an additional 3 Japanese patients aged 12 to 14 years will be enrolled to meet local regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply:

1. Parent(s)/guardian are able to give written informed consent prior to participation in the study, which will include the ability to comply with the requirements and restrictions listed in the consent form. If applicable, the participant must be able and willing to give assent to take part in the study according to the local requirement.
2. Patient must be 6 to 11 years of age inclusive (6 to 14 years of age inclusive in Japan), at the time of signing the ICF.
3. Diagnosis of severe asthma, defined by the regional guidelines for at least 12 months prior to Visit 1.
4. A previously confirmed history of two or more exacerbations requiring treatment with systemic corticosteroids and/or hospitalization in the 12 months prior to Visit 1.
5. Peripheral blood eosinophil count of ≥ 150 cells / µL at Visit 1.
6. A well-documented requirement for regular treatment with ICS: eg. total daily dose equivalent to ≥ 250 µg fluticasone propionate, in the 12 months prior to Visit 1, with or without maintenance oral corticosteroids.
7. Current treatment with at least 1 additional controller medication, such as inhaled LABA, leukotriene receptor antagonist, long acting anti-muscarinic agent, or theophylline, since at least 3 months prior to Visit 1.
8. Pre-bronchodilator FEV1 ≤ 110% predicted normal, or, FEV1/Forced Vital Capacity (FVC) ratio ≤ 0.8.
9. Body weight ≥15 kg.
10. Male or female
11. Females of childbearing potential (FOCBP) who are sexually active, as judged by the investigator, must commit to consistent and correct use of an acceptable method of contraception for the duration of the study and for 4 months after the last dose of IP.

Exclusion Criteria:

Patients are eligible to be included in the study only if all of the inclusion criteria and none of the exclusion criteria apply:

1. Any history of life-threatening asthma (eg, requiring intubation).
2. Clinically important pulmonary disease other than asthma such as active lung infection, bronchiectasis, pulmonary fibrosis, cystic fibrosis, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia.
3. Previous diagnosis of pulmonary or systematic disease, other than asthma, that is associated with elevated peripheral eosinophil counts such as allergic bronchopulmonary aspergillosis/mycosis, eosinophilic granulomatosis with polyangiitis (Churg-Strauss syndrome), and hypereosinophilic syndrome.
4. Ever been diagnosed with malignant disease.
5. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, immunological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

   1. Affect the safety of the patient throughout the study.
   2. Influence the findings of the study or their interpretations.
   3. Impede the patient's ability to complete the entire duration of the study.
6. History of anaphylaxis to any biologic therapy.
7. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the investigator may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete the entire duration of the study.
8. Any clinically significant cardiac disease or any electrocardiogram (ECG) abnormality obtained during the screening period, which in the opinion of the investigator may put the patient at risk or interfere with study assessments.
9. Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Patients with a history of hepatitis B vaccination without history of hepatitis B are allowed to enrol.
10. A helminth parasitic infection diagnosed within 24 weeks prior to the date of informed consent and assent is obtained that has not been treated with, or has failed to respond to, standard of care therapy.
11. Alanine aminotransferase or aspartate aminotransferase level ≥ 1.5 times the upper limit of normal confirmed during the screening period.
12. A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
13. Use of immunosuppressive medication, including, but not limited to, methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroid, or any experimental anti-inflammatory therapy, within 3 months prior to Visit 1. Chronic maintenance corticosteroid for the treatment of asthma is allowed.
14. Receipt of immunoglobulin or blood products within 30 days prior to Visit 1.
15. Receipt of any marketed (eg, Omalizumab, Mepolizumab, or off-label Benralizumab) or investigational biologic within 4 months or 5 half-lives, whichever is longer, prior to Visit 1.
16. Receipt of live attenuated vaccines 30 days prior to the date of first dose of IP.
17. Initiation of new allergen immunotherapy is not allowed within 30 days prior to Visit 1. However, allergen immunotherapy initiated prior to this period can be continued provided there is a gap of 7 days between the immunotherapy and IP administration.
18. Current use of any oral or ophthalmic non-selective β-adrenergic antagonist (eg, propranolol).
19. Planned surgical procedures during the conduct of the study.
20. Participation in another clinical study with an investigational nonbiologic product administered in the last 30 days or 5 half-lives prior to enrolment, whichever is longer.
21. Known history of allergy or reaction to any component of the IP formulation.
22. Concurrent enrolment in another clinical study.
23. Parent/guardian has a history of psychiatric disease, intellectual deficiency, substance abuse, or other condition (eg, inability to read, comprehend and write) which will limit the validity of consent to participate in this study.
24. Unwillingness or inability of the participant or parent/guardian to follow the procedures outlined in the protocol.
25. Children who are wards of the state or government.
26. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
27. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
28. Previous treatment in the present study.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Orlando, Florida
  - Research Site, Lincoln, Nebraska
  - Research Site, Cincinnati, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Coppell, Texas
  - Research Site, San Antonio, Texas
- Japan (7):
  - Research Site, Fukuoka
  - Research Site, Fukuyama-shi
  - Research Site, Gifu
  - Research Site, Habikino-shi
  - Research Site, Saga
  - Research Site, Tsu
  - Research Site, Zentsuji-shi

REFERENCES:
- [Derived] Wedner HJ, Fujisawa T, Guilbert TW, Ikeda M, Mehta V, Tam JS, Lukka PB, Asimus S, Durzynski T, Johnston J, White WI, Shah M, Werkstrom V, Jison ML; all TATE investigators. Benralizumab in children with severe eosinophilic asthma: Pharmacokinetics and long-term safety (TATE study). Pediatr Allergy Immunol. 2024 Mar;35(3):e14092. doi: 10.1111/pai.14092. PMID 38491795
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00025&attachmentIdentifier=293a579d-d532-4748-9486-04e94c6b2b6b&fileName=D3250C00025-clinical-study-report_synopsis_Redacted_PDFA.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, open-label, parallel group study was conducted in pediatric participants with severe eosinophilic asthma at 17 investigational sites in the United States and Japan between 21 Nov 2019 and 12 Sep 2022.
Pre-assignment Details: The study consisted of a screening period (up to 4 weeks), treatment period [2 parts; Part A (16 weeks) followed by Part B (32 weeks)], and a safety follow-up visit at Week 52.A total of 30 participants were enrolled in this study.
Groups:
- Benralizumab Dose 1, Aged 6-14 Years: All participants with body weight <35 kilograms (kg) at screening received benralizumab Dose 1 subcutaneous (SC) injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 1 at Weeks 24, 32, and 40 in Part B.
- Benralizumab Dose 2, Aged 6-14 Years: All participants with body weight >=35 kg or aged 12-14 years (irrespective of body weight) at screening received benralizumab Dose 2 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 2 at Weeks 24, 32, and 40 in Part B.
Period: Overall Study
Arm/Group | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Started | 15 | 15
Completed | 15 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by parent/guardian | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis set consisted of all participants who received at least 1 dose of benralizumab.
Groups:
- Benralizumab Dose 1, Aged 6-14 Years: All participants with body weight <35 kg at screening received benralizumab Dose 1 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 1 at Weeks 24, 32, and 40 in Part B.
- Total: Total of all reporting groups
Arm/Group | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (2.02) | 9.8 (1.93) | 9.0 (2.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 8
  Black or African American | 3 | 5 | 8
  Asian | 8 | 3 | 11
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Benralizumab
Description: Blood samples were collected to determine the clearance of benralizumab. This was an empirical Bayesian estimate (EBE) derived posthoc using population PK analysis.
Time Frame: Pre-dose on Days 0, 28, 56, 112, 168 and post-dose on Days 1, 7, 14, 84, 336; and at early discontinuation or withdrawal visit
Population: The PK analysis set consisted of all participants who received at least 1 dose of benralizumab for whom PK blood samples were not assumed to be affected by factors such as protocol violations and who had at least 1 post dose quantifiable serum PK observation.
Measure: Mean (Standard Deviation); unit: liter (L) per day
Groups:
- All Participants: All participants aged 6-14 years enrolled in this study irrespective of study treatment received were included in this arm.
Arm/Group | All Participants
Number analyzed (Participants) | 30
liter (L) per day | 0.156 (0.0598)

2. Primary Outcome: Area Under the Serum Concentration-Time Curve From Time Zero to Day 28 (AUC0-28) of Benralizumab
Description: Blood samples were collected to determine the AUC0-28 of benralizumab and it was calculated by linear up/log down trapezoidal summation. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Pre-dose on Days 0, 28 and post-dose on Days 1, 7, 14
Population: The Non-compartmental analysis (NCA) set consisted of all participants who received the first dose of benralizumab for whom PK blood samples were not assumed to be affected by factors such as protocol violations and who had at least 3 quantifiable serum PK observations post first dose on Days 1, 7, 14, and 28. Only those participants with data available were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*day per milliliter (ng*day/mL)
Groups:
- Benralizumab Dose 1, Aged 6-11 Years: Participants with body weight <35 kg at screening received benralizumab Dose 1 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 1 at Weeks 24, 32, and 40 in Part B.
- Benralizumab Dose 2, Aged 6-11 Years: Participants with body weight >=35 kg at screening received benralizumab Dose 2 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 2 at Weeks 24, 32, and 40 in Part B.
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 10 | 10 | 10 | 11
nanogram*day per milliliter (ng*day/mL) | 36918.01 (24.61) | 75593.37 (39.96) | 36918.01 (24.61) | 73670.51 (38.86)

3. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Benralizumab
Description: Blood samples were collected to determine Cmax of benralizumab and it was directly calculated from the individual concentration-time curve. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: as for outcome 1
Population: The NCA set consisted of all participants who received the first dose of benralizumab for whom PK blood samples were not assumed to be affected by factors such as protocol violations and who had at least 3 quantifiable serum PK observations post first dose on Days 1, 7, 14, and 28.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
ng/mL | 1901.18 (28.42) | 3118.69 (47.35) | 1901.18 (28.42) | 3090.85 (43.66)

4. Primary Outcome: Terminal Phase Elimination Half-Life (t1/2) of Benralizumab
Description: Blood samples were collected to determine the t1/2 of benralizumab and it was calculated as natural logarithm of 2 [ln(2)]/terminal rate constant (λZ). This was an EBE derived posthoc using population PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: day
Arm/Group | All Participants
Number analyzed (Participants) | 30
day | 14.4 [6.94 to 23.4]

5. Primary Outcome: Time to Achieve Maximum Observed Serum Concentration (Tmax) of Benralizumab
Description: Blood samples were collected to determine the tmax of benralizumab and it was directly calculated from the individual concentration-time curve. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: day
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
day | 6.91 [0.93 to 14.95] | 7.26 [1.10 to 14.01] | 6.91 [0.93 to 14.95] | 7.94 [1.10 to 14.01]

6. Primary Outcome: Trough Concentration of Benralizumab at Week 16 (Ctrough16)
Description: Blood samples were collected to determine the trough concentration at Week 16, the lowest concentration reached by benralizumab before the next dose was administered. The PK parameters were estimated using non-compartmental analysis method.
Time Frame: Pre-dose on Day 112
Population: The NCA set consisted of all participants who received the first dose of benralizumab for whom PK blood samples were not assumed to be affected by factors such as protocol violations and who had at least 3 quantifiable serum PK observations post first dose on Days 1, 7, 14, and 28. Only those participants with data available were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 14
ng/mL | 142.42 (256.34) | 339.35 (409.24) | 142.42 (256.34) | 340.46 (363.69)

7. Primary Outcome: Change From Baseline in Peripheral Blood Eosinophil Count up to Week 48
Description: Blood samples were collected for determination of eosinophil count levels and were assessed in a central laboratory. Baseline is the last non-missing measurement prior to the first dose of study treatment.
Time Frame: Baseline (Day 0) and at Weeks 4, 8, 12, 16, 24 and 48
Population: The Safety Analysis set consisted of all participants who received at least 1 dose of benralizumab. Only those participants with data available were analyzed.
Measure: Mean (Standard Deviation); unit: cells/microliters
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
cells/microliters
  Week 4 | -447.3 (283.76) | -436.9 (408.28) | -447.3 (283.76) | -455.3 (385.58)
  Week 8 | -445.3 (276.20) | -453.8 (396.03) | -445.3 (276.20) | -470.7 (374.25)
  Week 12: number analyzed (Participants) | 15 | 12 | 15 | 14
  Week 12 | -443.3 (286.85) | -455.8 (419.32) | -443.3 (286.85) | -472.9 (393.49)
  Week 16: number analyzed (Participants) | 15 | 11 | 15 | 12
  Week 16 | -446.7 (279.12) | -402.7 (384.61) | -446.7 (279.12) | -430.0 (378.68)
  Week 24: number analyzed (Participants) | 12 | 13 | 12 | 14
  Week 24 | -354.2 (323.99) | -436.9 (405.90) | -354.2 (323.99) | -457.9 (397.77)
  Week 48: number analyzed (Participants) | 15 | 13 | 15 | 14
  Week 48 | -434.0 (286.15) | -453.8 (392.78) | -434.0 (286.15) | -474.3 (385.04)

8. Secondary Outcome: Body Weight-Adjusted Clearance of Benralizumab
Description: Blood samples were collected to determine the clearance of benralizumab. This was an EBE derived posthoc using population PK analysis.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/day/kilogram
Arm/Group | All Participants
Number analyzed (Participants) | 30
L/day/kilogram | 0.00408 (0.000764)

9. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Response to Benralizumab
Description: Blood samples were analyzed for the presence of ADAs for benralizumab. ADA prevalence: ADA positive (+ve) at any time point including baseline and/or post baseline. Treatment induced ADA+ve: ADA negative (-ve) at baseline and post-baseline ADA+ve. Treatment-boosted ADA+ve: baseline +ve ADA titer that was boosted by >4-fold or higher-level following study drug administration. Treatment-emergent ADA+ve: either treatment-induced ADA+ve or treatment-boosted ADA+ve. Persistently +ve ADA: having at least 2 post-baseline ADA+ve assessments with at least 16 weeks (112 days) between the first and last +ve assessments, or an ADA+ve result at the last available assessment. Transiently +ve ADA: having at least 1 post-baseline ADA+ve assessment(s) and not persistently ADA+ve. Neutralizing antibodies (nAb) prevalence: nAb+ve at baseline and/or post-baseline. Treatment-induced nAb+ve (nAb incidence): nAb-ve at baseline (or ADA-ve at baseline) and nAb+ve at any post-baseline visit.
Time Frame: Pre-dose at Baseline (Day 0), Weeks 8, 16 and 24 and post-dose at Week 48; and at early discontinuation or withdrawal visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
Participants
  ADA prevalence | 3 | 1 | 3 | 1
  Treatment-emergent ADA+ve | 3 | 1 | 3 | 1
  Post-baseline ADA+ve | 3 | 1 | 3 | 1
  Baseline and at least 1 post-baseline ADA+ve: number analyzed (Participants) | 13 | 13 | 13 | 15
  Baseline and at least 1 post-baseline ADA+ve | 0 | 0 | 0 | 0
  Only baseline ADA+ve: number analyzed (Participants) | 13 | 13 | 13 | 15
  Only baseline ADA+ve | 0 | 0 | 0 | 0
  Persistently ADA+ve | 1 | 0 | 1 | 0
  Transiently ADA+ve | 2 | 1 | 2 | 1
  nAb prevalence | 3 | 1 | 3 | 1
  nAb incidence | 3 | 1 | 3 | 1

10. Secondary Outcome: Change From Baseline in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) up to Week 48
Description: The FEV1 was defined as the volume of air exhaled from the lungs in the first second of a forced expiration and was measured by spirometry. Baseline is the last non-missing measurement with acceptable quality prior to the first dose of study treatment.
Time Frame: Baseline (Day 0) and at Weeks 16 and 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
liters
  Week 16: number analyzed (Participants) | 11 | 7 | 11 | 8
  Week 16 | -0.001 (0.2434) | -0.119 (0.2435) | -0.001 (0.2434) | -0.165 (0.2609)
  Week 48: number analyzed (Participants) | 15 | 12 | 15 | 13
  Week 48 | 0.003 (0.3412) | 0.425 (0.4395) | 0.003 (0.3412) | 0.428 (0.4209)

11. Secondary Outcome: Change From Baseline in Interviewer-Administered Asthma Control Questionnaire (ACQ-IA) Score up to Week 48
Description: The ACQ-IA is a 6-item assessment comprised of 6 patient-reported items. Participants were asked to record their experience with 5 symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, and wheezing) and use of short-acting beta-2 agonist (SABA) over the previous week using a 7-point scale (0 = no impairment; and 6 = maximum impairment). The ACQ-IA score was calculated by the mean of the 7 equally weighted items. The score ranged from 0 (well controlled) to 6 (extremely poorly controlled). Higher scores indicated poor asthma control. Baseline is the last non-missing measurement prior to the first dose of study treatment.
Time Frame: Baseline (Day 0), at Weeks 16 and 48; and at early discontinuation or withdrawal visit
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
scores on a scale
  Week 16: number analyzed (Participants) | 15 | 12 | 15 | 13
  Week 16 | -0.62 (0.890) | -1.18 (1.717) | -0.62 (0.890) | -1.06 (1.696)
  Week 48: number analyzed (Participants) | 14 | 12 | 14 | 13
  Week 48 | -0.56 (1.252) | -1.36 (1.369) | -0.56 (1.252) | -1.31 (1.324)

12. Secondary Outcome: Number of Responders in Interviewer-Administered Patient Global Impression of Change (PGIC)-IA and Clinician Global Impression of Change (CGIC) Questionnaires
Description: The PGIC-IA and CGIC instruments were used for an overall evaluation of response to treatment, conducted separately by the Investigator and by the participant (administered by trained individuals to help the child understand the question and response options), using a 7-point scale: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; and 7=very much worse. The Investigator (clinician) and the participant were asked to rate the degree of change in the overall asthma status compared to the start of study treatment visit. Participants were defined as responders based on categorized responses for PGIC-IA and CGIC. Responder status categories included Improved=Very much improved, Much improved, Minimally improved, Much improved=Much improved, Very much improved, Very much improved=Very much improved. CGIC = PGIC-IA indicates agreement between CGIC and PGIC-IA assessments of response to treatment at the same visit.
Time Frame: At Weeks 16 and 48; and at early discontinuation or withdrawal visit
Population: The Safety Analysis set consisted of all participants who received at least 1 dose of benralizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
Number analyzed (Participants) | 15 | 13 | 15 | 15
Participants
  PGIC-IA, Week 16, improved | 13 | 12 | 13 | 13
  PGIC-IA, Week 16, much improved | 10 | 10 | 10 | 11
  PGIC-IA, Week 16, very much improved | 4 | 8 | 4 | 9
  PGIC-IA, Week 48, improved | 13 | 12 | 13 | 13
  PGIC-IA, Week 48, much improved | 9 | 10 | 9 | 11
  PGIC-IA, Week 48, very much improved | 9 | 9 | 9 | 10
  CGIC, Week 16, improved | 13 | 11 | 13 | 12
  CGIC, Week 16, much improved | 8 | 9 | 8 | 9
  CGIC, Week 16, very much improved | 3 | 5 | 3 | 5
  CGIC, Week 48, improved | 15 | 13 | 15 | 14
  CGIC, Week 48, much improved | 8 | 11 | 8 | 12
  CGIC, Week 48, very much improved | 5 | 6 | 5 | 6
  CGIC = PGIC-IA, Week 16, improved | 10 | 6 | 10 | 6
  CGIC = PGIC-IA, Week 16, much improved | 7 | 5 | 7 | 5
  CGIC = PGIC-IA, Week 16, very much improved | 3 | 4 | 3 | 4
  CGIC = PGIC-IA, Week 48, improved | 9 | 8 | 9 | 8
  CGIC = PGIC-IA, Week 48, much improved | 5 | 7 | 5 | 7
  CGIC = PGIC-IA, Week 48, very much improved | 5 | 6 | 5 | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of study drug administration (Day 1) until end of follow-up, approximately up to Week 53
Description: The Safety Analysis set consisted of all participants who received at least 1 dose of benralizumab.
Groups:
- Benralizumab Dose 1, Aged 6-14 Years: All participants with a body weight <35 kg at screening received benralizumab Dose 1 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 1 at Weeks 24, 32, and 40 in Part B.
- Benralizumab Dose 2, Aged 6-14 Years: All participants with a body weight >=35 kg or aged 12-14 years (irrespective of body weight) at screening received benralizumab Dose 2 SC injection once daily on Day 0 and at Weeks 4, 8, and 16 in Part A, followed by benralizumab Dose 2 at Weeks 24, 32, and 40 in Part B.
Arm/Group | Benralizumab Dose 1, Aged 6-11 Years | Benralizumab Dose 2, Aged 6-11 Years | Benralizumab Dose 1, Aged 6-14 Years | Benralizumab Dose 2, Aged 6-14 Years
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/13 | 1/15 | 4/15
Other Adverse Events (participants affected / at risk) | 13/15 | 9/13 | 13/15 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab Dose 1, Aged 6-11 Years (N=15) | Benralizumab Dose 2, Aged 6-11 Years (N=13) | Benralizumab Dose 1, Aged 6-14 Years (N=15) | Benralizumab Dose 2, Aged 6-14 Years (N=15)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab Dose 1, Aged 6-11 Years (N=15) | Benralizumab Dose 2, Aged 6-11 Years (N=13) | Benralizumab Dose 1, Aged 6-14 Years (N=15) | Benralizumab Dose 2, Aged 6-14 Years (N=15)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1) | 3 (4) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Allergy to animal (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Immunisation reaction (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (5) | 1 (1) | 4 (5) | 2 (3)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (3) | 2 (2) | 2 (3)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occult blood positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (4) | 1 (1) | 2 (4) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (3) | 0 (0) | 1 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04305405/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT04305405/SAP_001.pdf